CLINICAL TRIAL: NCT04010279
Title: The Effects of Setting Adjustable Pressure Limiting Valve (APL) to 5 cmH2O on Preoxygenation
Brief Title: Can we Improve Preoxygenation by Using Adjustable Pressure Limiting Valve (APL) ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, MAHMUT ARSLAN, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KSU 2019-77
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Preoxygenation
Keywords: preoxygenation; CPAP(continuous positive airway pressure); APL (airway pressure release) valve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- spontaneous breathing (Active Comparator): volunteers will breath via an anesthesia face mask spontaneously while the APL (airway pressure release valve) valve is on the spontaneous position.
  Interventions: Procedure: preoxygenation with 100% O2, fresh gas flow rate 12 L/minute
- spontaneous breathing with APL 5 cmH2O (Active Comparator): volunteers will breath via an anesthesia face mask spontaneously while the APL (airway pressure release valve) valve is on the 5 cmH2O position.
  Interventions: Procedure: preoxygenation with 100% O2, fresh gas flow rate 12 L/minute
- CPAP 5cmH2O PEEP (Active Comparator): volunteers will breath via an anesthesia face mask spontaneously on the CPAP mode of the anesthesia workstation with 5 cmH2O PEEP.
  Interventions: Procedure: preoxygenation with 100% O2, fresh gas flow rate 12 L/minute

INTERVENTIONS:
Procedure: preoxygenation with 100% O2, fresh gas flow rate 12 L/minute — volunteers will be placed in supine position, fresh gas flow rate will be set at 12 L/min and delivered oxygen concentration will be set at 100%.

SUMMARY:
The aim of this study is to investigate the effects of setting airway pressure release valve (APL valve) on the anesthesia workstation to 5 cmH2O during spontaneous breathing on preoxygenation. In this prospective study healthy volunteers are randomized in cross-over between spontaneous breathing with the APL valve on spontaneous position or spontaneous breathing with the APL valve on 5 cmH2O or CPAP (continous positive airway pressure) mode with 5 cmH2O PEEP (positive end expiratory pressure).

DETAILED DESCRIPTION:
There are several methods to improve preoxygenation but most of them require advanced anesthesia workstations. Therefore the investigators planned an an experimental study on healthy volunteers to investigate the effects of a simple method on preoxygenation.

Healthy volunteers are randomized in cross-over between spontaneous breathing with the APL valve on spontaneous position or spontaneous breathing with the APL valve on 5 cmH2O or CPAP mode with 5 cmH2O PEEP.

The volunteers will breath through an anesthesia face mask. The fresh gas flow rate is 12 L/min, inspiratory fraction of oxygen is 100%. The exhaled gas (oxygen and carbon dioxide) are monitored. The inspiratory and end expiratory fraction of oxygen will be recorded every 10 seconds.

The primary endpoint is the time to achieve end expiratory fraction of oxygen of 90% or more.The secondary endpoint is the proportion of subject with end expiratory fraction of oxygen of 90% or more after a 3 min period and the end expiratory fraction of oxygen at the third minute.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any respiratory disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
time to reach end expiratory fraction of oxygen of 90% or more | 5 minutes

SECONDARY OUTCOMES:
proportion of volunteer with end expiratory fraction of oxygen of 90% or more after a 3 min period | 3 minutes
End expiratory oxygen fraction at the 3th minute | 3 minutes
Verbal rating Score | 5 minutes
  After completion of the whole arms of the study the volunteers will give a score between 0-10 to define the difficulty of breathing during the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş, In the USA Or Canada, Please Select...
  - KAhramanmaras Sutcu Imam University, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hanouz JL, Le Gall F, Gerard JL, Terzi N, Normand H. Non-invasive positive-pressure ventilation with positive end-expiratory pressure counteracts inward air leaks during preoxygenation: a randomised crossover controlled study in healthy volunteers. Br J Anaesth. 2018 Apr;120(4):868-873. doi: 10.1016/j.bja.2017.12.002. Epub 2018 Jan 17. PMID 29576128
- [Result] Sreejit MS, Ramkumar V. Effect of positive airway pressure during pre-oxygenation and induction of anaesthesia upon safe duration of apnoea. Indian J Anaesth. 2015 Apr;59(4):216-21. doi: 10.4103/0019-5049.154998. PMID 25937647